CLINICAL TRIAL: NCT01044121
Title: A Latin-Square Crossover Study of the Effects of Mattress Firmness on Pain in Patients With Chronic Low-Back Pain
Brief Title: Effects of Mattress Firmness on Pain in Patients With Chronic Low-Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sleep To Live Institute (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Duke-Pain-1113291
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Low Back Pain; Sleep Disruption
Keywords: mattress; pain; sleep; low back pain; back; neck; arousal; pillow; kingsdown; sleep to live; duke university; sleep to live institute; missouri; springfield; joplin; body diagnostic; dormo diagnostic; morning pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Mattress Firmness (Experimental)
  Interventions: Other: Mattress Firmness

INTERVENTIONS:
Other: Mattress Firmness — Current mattress and 6 experimental firmnesses of mattress as defined by a Comfort Support Analysis device.
  Other Names: Kingsdown; Sleep to Live

SUMMARY:
The primary study objective is to determine whether mattress firmness affects pain in patients with chronic low-back pain. We hypothesize that mattresses that differ in their firmness and support should have a varying effect on low-back pain patients' level of pain and pain-related disability. We also seek to test the hypothesis that the optimal mattress might vary from person to person.

In this regard, we will test:

1. Whether there is a single mattress that is superior to the others in terms of reducing low-back pain and pain related disability.
2. Whether the optimal mattress for reducing pain varies in the observed population.

DETAILED DESCRIPTION:
Few treatments are effective for chronic low-back pain, a disorder that causes marked social costs in developed countries. A "comfortable" mattress is commonly assumed to play an essential role, both on a preventive and on a therapeutic basis on chronic low-back pain. However, evidence supporting the beneficial effects of different levels of mattress support on pain is lacking.

The primary study objective is to determine whether mattress firmness affects pain in patients with chronic low-back pain. We hypothesize that mattresses that differ in their firmness and support should have a varying effects on LBP patients' level of pain and pain-related disability. We also seek to test the hypothesis that the optimal mattress might vary from person to person. In this regard, we will test:

1. whether there is a single mattress that is superior to the others in terms of reducing low-back pain and pain-related disability and
2. whether the optimal mattress for reducing pain varies in the observed population.

The secondary objectives are:

1. to determine whether there is a relationship between mattress firmness and sleep in this population;
2. to determine whether there is a relationship between pain and sleep in this population;
3. to determine whether key sleep variables (subjective or objective) are mediating or moderating factors of the relationship between mattress and level of low-back pain (LBP) and disability;
4. to determine if different sleep surfaces have differential effects on measures of daily function among patients with chronic LBP;
5. to evaluate if Kingsdown's proprietary algorithm for selecting optimal mattress "fits" with the subject's best mattress for reducing pain and improving sleep and measures of daytime functioning;
6. to conduct exploratory regression analyses using variables included in the proprietary algorithm and other demographics and measures of physical characteristics to predict the optimal "fit" mattress (i.e., the mattress associated with lowest morning pain ratings, best sleep measures and optimal levels of daytime function);
7. to determine if different sleep surfaces have differential effects on measures of partner sleep disturbance;
8. to determine if there is a relationship between partner pain level and partner sleep disturbances.

Please see "Eligibility Criteria" for inclusion and exclusion information.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain location must be inferior to T12 and superior to the gluteal fold and chronic (greater than 3 months)
* Patient Global Impression for Pain of at least 3 on a 1-5 scale (moderate severity)
* Visual Analog Scale for Pain of at least 40 on a 100 point scale (0 = no pain; 100 = worst pain)
* Presence of normal motor strength on exam
* English speaking and reading man/woman between the ages of 21-64

Exclusion Criteria:

* Neurologic or medical illness that is directly responsible for back pain
* Psychiatric disease
* Back related surgery
* Substance abuse
* Pregnancy (self or partner)
* Sleep-affecting medications
* Recent surgery
* Recent physical trauma
* Fibromyalgia
* Spinal Stenosis
* Sciatica
* Spondylolisthesis
* Spondyloarthropathy
* Sciatica
* Spinal Stenosis
* Vertebral Fractures
* Rheumatoid Arthritis
* Inability to comply
* Untreated sleep disorders
* Night-shift worker
* Frequent travel
* Parent of child under 2
* Pending litigation for pain issue
* Corticosteroid use in the last 90 days

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Reduction of Pain | Daily and every 3 weeks

SECONDARY OUTCOMES:
Improved Sleep Quality | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Robert Oexman, DC, Principal Investigator — Sleep To Live Institute